CLINICAL TRIAL: NCT05872165
Title: Influence Of Ozonated Gel Phonophoresis In The Treatment Of Chronic Lateral Epicondylitis
Brief Title: Ozonated Gel Phonophoresis On Chronic Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Elaziz Mohamed Hefny, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of cairo PHT
Record Dates: First submitted 2023-05-12; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Epicondylitis
MeSH Terms: interventions — Phonophoresis; Ultrasonography; Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): this group of 20 subjects will receive the ozonated media phonophoresis plus conventional physical therapy program 3 times weekly for 4 weeks.
  Interventions: Device: phonophoresis; Other: conventional physical therapy
- Control group (Other): this group of 20 subjects will receive only conventional physical therapy program 3 times weekly for 4 weeks.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Device: phonophoresis — 1 MHz, 1 W/cm2continuous mode of ultrasound therapy for 5 min. using ozonated gel as a coupling medium
  Other Names: Ultrasound with ozonated medium gel
  Arms: Experimental group
Other: conventional physical therapy — conventional TENS (100 Hz) for 30 min - hot pack for 20 min- stretching and strengthening exercises, wrist rest splints 3times per week for 4 weeks.
  Other Names: Tens and exercises

SUMMARY:
Comparison between 2 groups of chronic lateral epicondylitis, to determine the effect of ozonated media phonophoresis on chronic lateral epicondylitis.

DETAILED DESCRIPTION:
40 patients (male and female), patients age would be ranged from 30 to 50 years, would be randomly allocated using sealed envelope into randomly two matched group (A and B), Group A (Experimental): 20 patients would receive ultrasonic with ozonated gel as a coupling medium (phonophoresis) (1 MHz, 1 W/cm2continuous mode) for 5 min. plus, conventional physical therapy program consists of (conventional TENS (100 Hz) for 30 min - hot pack for 20 min- stretching and strengthening exercises, wrist rest splints). 3 times per week for 4 weeks.

Group B (control):20 patients will receive conventional physical therapy program consists of (conventional TENS (100 Hz) for 30 min - hot pack for 20 min- stretching and strengthening exercises, wrist rest splints) 3times per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients would be diagnosed as chronic lateral epicondylitis from both genders.
* Patients with chronic lateral epicondylitis that diagnosed by orthopedist.
* Positive clinical manifestation in all patients.
* Pain onset is more than 3 months.
* All participants must be medically stable and not be treated with analgesics or any medication which may cause misleading results.
* All patients had body mass index between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

* Subjects would be excluded if they have:

Received intra articular injection from duration less than 3 months.

* Elbow instability.
* History of cancer.
* Pregnancy
* Infection.
* Skin diseases on elbow area.
* Open wound in elbow.
* Shoulder or elbow fractures
* Systemic diseases such as rheumatoid arthritis, Reiter's syndrome, or diabetes.
* Neurological diseases.
* Severe medical or psychiatric disorders.
* Elbow surgery.
* Entrapment of the radial nerve.
* Arthritis and effusion of the elbow.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain status | 4 weeks
  assessment of pain using (visual analogue scale)s a horizontal line, 100 mm in length, anchored by word descriptors at each end. 2) The patient mark millimeters ed on the line the point that they feel ed represents their perception of their current state. The VAS score is determined by measuring in from the start point of the line to the point that the patient marks It was used to evaluate pain intensity. The VAS is a self. reported pain meas urement scale. The extremes of the line are labelled as no pain and worst pain. Each subject was asked to mark the point on the line that exactly corresponded to his/her pain .
wrist ROM | 4 weeks
  Measurment of wrist range of motion using universal goniometer
Hand grip strength | 4 weeks
  measurment of hand grip strength using hand grip dynamometer

IPD SHARING:
Plan to Share IPD: No
think to share after request.